CLINICAL TRIAL: NCT04430205
Title: Repair of Vertically Fractured Root: An Observational Clinical Study
Brief Title: Repair of Vertically Fractured Root
Status: Completed | Type: Observational
Sponsor: Centro di Ricerca Odonotiatrica e Corsi di Aggiornamento Professionale (Other)
Responsible Party: Principal Investigator, Fabrizio Zaccheo, Principal Investigator, Centro di Ricerca Odonotiatrica e Corsi di Aggiornamento Professionale
Other Study IDs: 2370CELazio1
Record Dates: First submitted 2020-06-05; First posted 2020-06-12 (Actual); Last update posted 2020-06-12 (Actual); Status verified 2020-06

CONDITIONS: Root; Fracture
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Adhesive restoration protocol — The canal walls were etched with 37% orthophosphoric acid for 30 seconds with use of a microbrush.
  The primer was applied on the wet canal walls, with a microbrush several times, after checking by drying the canal, that the appearance of the dentine was shiny and not opaque or chalky.
  The next step was the application of bonding with a microbrush, blowing in the fracture line to make sure it is not loaded with bonding.
  Flow composite was used to make it penetrate the fracture line with the help of a 0.06 mm k-file.
  The canals were filled with dual composite parts more deeply, light cured at the canal entrance and pulp chamber; the following phase was the coronal restoration with a sandwich technique, covering the cusp with composite.

SUMMARY:
Aim and background: The aim of this retrospective observational study is to evaluate the survival rate of cracked teeth, presenting partial (PVF) or complete vertical fracture (CVF), after tooth restoration either with fracture-fragment adhesive bonding or with amalgam restoration.

Materials and Methods: One hundred eight fractured teeth, from 99 patients (51 males, 48 females, mean age 50.5 years), presenting complete or partial root fracture, were treated with adhesive restoration or non-adhesive restoration protocol (amalgam) between 1991 and 2019. Demographic and clinical variables were evaluated as predictors of extraction. Furthermore, the bone loss/recovery due to therapy for the fracture was radiographically evaluated at the one year follow-up. All cases were treated by the same operator, using a surgical microscope. Statistical analysis was performed with IBM SPSS Statistics. The study was approved by the ethical committee of Sistema Sanitario Nazionale (prot. N°2370CELazio1).

DETAILED DESCRIPTION:
One hundred eight fractured teeth, from 99 patients (51 males, 48 females, mean age 50.5 years, standard deviation (SD) 12.8, range 23-84), presenting complete or partial root fracture, were included in this observational retrospective study. All the teeth were treated according to one of two clinical protocols (adhesive or amalgam, see below). Besides a general medical history and subjective and objective symptoms, the presence of the crack was determined by the usage of a Leica 650 stereomicroscope with the help of methylene blue or eosin-type dyes. The following parameters were gathered from the clinical charts to evaluate possible risk factors for extraction: age, gender, tooth number and type of root fracture (complete or partial). A vitality test was performed with an electrical test, and periodontal probing was performed on six sites per tooth to detect probing defects, using a manual probe. Periapical radiolucency at the moment of the diagnosis, survival in months and type of coronal restoration at the diagnosis (no restoration, single crown, composite, amalgam) were all explored. Presence of calcification in the canal, endo-treatment before the diagnosis of fracture (no treatment, good endodontic treatment, surgical treatment, retreatment), canal obstacles (i.e., broken files) and previous endo-canal retention (no retention, screw post, fibre post, cast post, composite, amalgam) were all determined. Survival was also considered at one, three, five and more than five years, and a qualitative evaluation of the tooth was given (success, functional success: the tooth was asymptomatic; failure: the tooth would be extracted; extracted: the tooth was extracted before the control visit), modifying the European Society of Endodontology for success of endodontic therapies. When evaluating treatment results, a commission made up of three operators, all active members of the Italian Endodontic Society (SIE), re-examined the radiograms and the clinical chart.

The bone loss/recovery due to the therapy of the fracture was radiographically evaluated at the one year follow-up: using Adobe Photoshop, the area of the bone loss was drawn, calculated and compared on radiograms at the moment of the diagnosis and at one year after the treatment, using the same radiological projection and classified as recovered, same loss, or further loss.

Radiographic examination was performed after the restoration, and then the radiographic survey was repeated every six months for the first two years and once a year for the remaining period.

These cases have all been reported, treated and evaluated over time by radiographic and clinical investigation. In all treated cases, the protocol of adhesive restorations was the same, performed and documented with the aid of the Leica 650 surgical microscope by the same operator. The adhesive protocol (87 cases) remained unchanged over time (from 1991 to 2019). A few cases (21 cases) were treated with amalgam, following protocols recommended by the literature to avoid the risk of dental fractures (endo-canal retention and cusp covering).

ELIGIBILITY:
Inclusion Criteria:

Any patient with at least one tooth with a vertical root fracture

Exclusion Criteria:

any patient who does not have at least one tooth with a vertical root fracture

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: One hundred eight fractured teeth, from 99 patients (51 males, 48 females, mean age 50.5 years, standard deviation (SD) 12.8, range 23-84), presenting complete or partial root fracture
Sampling Method: Non-Probability Sample
Enrollment: 99 (Actual)
Dates: Start 1991-07-15 (Actual); Primary Completion 2019-09-05 (Actual); Study Completion 2019-12-19 (Actual)

PRIMARY OUTCOMES:
Results | from 1991 to 2019
  Survival rate of teeth with vertical root fracture will be considered at one, three, five and more than five years, and a qualitative evaluation of the tooth will be given, clinically and radiographically:
  * success: tooth is asymptomatic and there is not radiographc lesion;
  * functional success: the tooth is asymptomatic but there is a radiographic lesion;
  * failure: the tooth would be extracted because of symptoms and/or radiographic lesion getting worse;
  * extracted: the tooth was extracted before the control visit.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Malentacca A, Zaccheo F, Scialanca M, Fordellone F, Rupe C, Lajolo C. Repair of teeth with cracks in crowns and roots: An observational clinical study. Int Endod J. 2021 Oct;54(10):1738-1753. doi: 10.1111/iej.13598. Epub 2021 Aug 16. PMID 34291470